CLINICAL TRIAL: NCT04591093
Title: Study of Musical Perception and Post-operative Auditory Performance as a Function of the Depth of Stimulation in Subjects Implanted With a MED-EL Cochlear Implant and Using a FineHearing Strategy Single-center Randomized Cross-over Study
Brief Title: Auditory Performances With Different Stimulation Depths in Cochlear Implanted Subjects Using a Fine Structure Strategy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MED-EL_FS_stimdepth_frenchstud
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant; stimulation strategy; sound coding strategy
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Crossover Assignment two arms A and B: Arm A: patient's fitting with strategy FS4 and 10 more apical electrodes activated--> 1 month use --> tests and patient's fitting with strategy FS4 and 10 more basal electrodes --> 1 month use --> tests
  Arm B: patient's fitting with strategy FS4 and 10 more basal electrodes activated --> 1 month use --> tests and patient's fitting with strategy FS4 and 10 more apical electrodes --> 1 month use --> tests
Who Masked: Participant, Investigator
Masking Description: Double blind study: the patient and the investigator don't know the strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CI with FineHearing with 10 more apical electrodes activated then 10 more basal electrodes activated (Active Comparator): Cochlear implant with FineHearing Strategy with 10 more apical electrodes activated first during 1 month then FineHearing Strategy with 10 more basal electrodes activated during 1 month
  Interventions: Device: FineHearing Strategy with 10 more apical electrodes or with 10 more basal electrodes activated
- CI with FineHearing with 10 more basal electrodes activated then 10 more apical electrodes activated (Active Comparator): Cochlear implant with FineHearing Strategy with 10 more basal electrodes activated first during 1 month then FineHearing Strategy with 10 more apical electrodes activated during 1 month
  Interventions: Device: FineHearing Strategy with 10 more apical electrodes or with 10 more basal electrodes activated

INTERVENTIONS:
Device: FineHearing Strategy with 10 more apical electrodes or with 10 more basal electrodes activated — Cochlear implant with FineHearing Strategy with 10 more apical electrodes activated or with 10 more basal electrodes activated

SUMMARY:
Main objective:

Investigate on new cochlear implanted patients whether the FineHearing strategy of the MED-EL cochlear implant gives better results on musical perception if the depth of stimulation (stimulation or not of the apical areas) is greater.

Secondary objectives:

Evaluate the effect of stimulation depth on vocal audiometric results, results of differential frequency threshold test and on qualitative sound perception.

DETAILED DESCRIPTION:
Introduction:

Conventional stimulation strategies in cochlear implants (e.g. ACE, CIS) use the place of the electrode to code the frequency by sending low frequency information on the apical electrodes and high frequency information on the basal electrodes. The stimulation rate of the electrodes is constant.

The pitch is only partially transmitted by these conventional strategies which would explain the poor results of cochlear implants in the perception of music.

In the FineHearing strategy of the MED-EL implant, the rate of stimulation on the low-frequency electrodes is related to the frequency of the sound and makes it possible to code the frequency information temporally.

Rader & al. 2016 have studied the contribution of adding to the tonotopic coding of the frequency (classical strategy) a temporal coding of the information by varying the stimulation rate. The results obtained show that providing this frequency information by time coding makes it possible to obtain perceived pitch much closer to the expected pitch (of normal-hearing) and less variability, especially at low frequencies. With fixed stimulation rate (classical strategy) low frequencies are poorly coded, whereas with the variable stimulation rate they are better coded.

In addition, Landsberger et al. [2018] studied in six subjects with a MED-EL implant the perception of a temporal coding according to the position of the electrodes with a long insertion: middle or apical position. The results seem to show that the temporal coding of the frequency would be more reliable than the spatial coding (related to the position of the electrode) at the apex, and the reverse on the electrodes in the middle position.

Studies have shown that the FineHearing strategy can provide benefits over the classic HDCIS strategy in tasks involving the fundamental F0 such as speech recognition in noise (after a certain learning time) [Kleine Punte & al. 2014 ; Vermeire & al. 2010], the perception of music [Roy & al. 2015 ; Roy & al. 2016] or the perceived quality of pitch [Müller & al. 2012].

The results obtained seem to depend on the position of the electrode: a deep insertion to reach the apical zone of the cochlea would allow better coding of the information.

MED-EL's FineHearing coding strategy with stimulation of the apical areas of the cochlea (long insertion of electrodes) could therefore allow better transmission of musical pitch and in particular improve the subjective quality of music compared to the same stimulation strategy without reaching the apical areas (short insertion).

Objective of the study: The objective of the study is to evaluate if the FineHearing strategy of MED-EL with stimulation of the apical zones allows to better transmit musical pitch and in particular to improve the subjective quality of the music compared to the same stimulation strategy without apical stimulation.

Main objective:

Show that the FineHearing strategy of MED-EL with stimulation of the apical zones allows to obtain a better perceptual quality of music in newly implanted cochlear patients than the same strategy without apical stimulation.

Secondary objectives:

* Evaluate differential frequency thresholds and correlation with qualitative perceptions of music.
* Evaluate the effect of the stimulation of the apical zones on the results of speech audiometry with the FineHearing strategy.
* Evaluate the effect of the stimulation of the apical zones on the subjective quality of sounds by questionnaire with the FineHearing strategy.

Plan of study:

it is a Single-center, randomized, double-blind, cross-over study

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation
* Patient with a postoperative insertion angle of the apical electrode > 450°
* Patient with 12 active electrodes on the day of activation.

Exclusion Criteria:

* Retro-cochlear pathology: auditory neuropathy, vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative measure of music with direct audio link | at 1 month post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sounds, loudness.
  Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).
  The test is performed with a direct audio link to the CI.
Qualitative measure of music with direct audio link | at 2 months post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sounds, loudness.
  Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).
  The test is performed with a direct audio link to the CI.

SECONDARY OUTCOMES:
Qualitative measure of music | at 1 month post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sounds, loudness.
  Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).
  The test is performed in free field without any contralateral aid.
Qualitative measure of music | at 2 months post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sounds, loudness.
  Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).
  The test is performed in free field without any contralateral aid.
Speech recognition in quiet | at 1 month post-activation
  The speech recognition in quiet is evaluated with 3 monosyllabic list of 17 words at 60 dB SPL. The patient has to recognize 17 words and 51 phonemes. The words and phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 for the words and the phonemes (or 0% and 100%).
Speech recognition in quiet | at 2 months post-activation
  The speech recognition in quiet is evaluated with 3 monosyllabic list of 17 words at 60 dB SPL. The patient has to recognize 17 words and 51 phonemes. The words and phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 for the words and the phonemes (or 0% and 100%).
Differential frequency threshold | at 1 month post-activation
  This test aimed to determine the smallest perceptible difference in F0 between two stimuli for various baseline values of F0. An adaptive procedure is used.
Differential frequency threshold | at 2 months post-activation
  This test aimed to determine the smallest perceptible difference in F0 between two stimuli for various baseline values of F0. An adaptive procedure is used.
Sound quality | at 1 month post-activation
  The HISQUI questionnaire will be used to evaluate the sound quality. The HISQUI questionnaire (Hearing Implant Sound Quality Index) is a questionnaire on the perceptual quality of sounds given a score (maximum=203) for each patient which indicates how he/she perceives the sound quality with his/her hearing implant in the everyday life.
Sound quality | at 2 months post-activation
  The HISQUI questionnaire will be used to evaluate the sound quality. The HISQUI questionnaire (Hearing Implant Sound Quality Index) is a questionnaire on the perceptual quality of sounds given a score (maximum=203) for each patient which indicates how he/she perceives the sound quality with his/her hearing implant in the everyday life.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mosnier, Dr, Principal Investigator — Service ORL, UF Implants auditifs et explorations fonctionnelles GH Pitié-Salpêtrière, APHP 6 Paris
Locations (1):
- GH Pitié-Salpêtrière, APHP 6, Paris, France